CLINICAL TRIAL: NCT01742572
Title: NEW Dietary Interventions to Enhance the Treatments for Weight Loss (NEW DIETs for Weight Loss Study)
Brief Title: New DIETs: New Dietary Interventions Enhancing the Treatment for Weight Loss
Acronym: New DIETs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Brie Turner-McGrievy, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00021116
Record Dates: First submitted 2012-11-27; First posted 2012-12-05 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Overweight; Obesity
Keywords: weight loss; obesity; overweight; diet
MeSH Terms: conditions — Overweight; Obesity; Weight Loss | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Vegan (Experimental): A vegan diet is one that does not contain any animal products (no meat, fish, poultry, eggs, or dairy) but emphasizes plant-based foods, such as fruits, vegetables, whole grains, and legumes/beans. We will also ask you to keep foods low in fat and low in glycemic index.
  Interventions: Behavioral: Diet
- Vegetarian (Experimental): A vegetarian diet is one that does not contain meat, fish, or poultry but does contain eggs and dairy, in addition to plant-based foods, such as fruits, vegetables, whole grains, and legumes/beans. We will also ask you to keep foods low in fat and low in glycemic index.
  Interventions: Behavioral: Diet
- Pesco-Vegetarian (Experimental): A pesco-vegetarian diet is one that does not contain meat or poultry but does contain fish and shellfish, eggs, and dairy, in addition to plant-based foods, such as fruits, vegetables, whole grains, and legumes/beans. We will also ask you to keep foods low in fat and low in glycemic index.
  Interventions: Behavioral: Diet
- Semi-Vegetarian (Experimental): A semi-vegetarian diet is one that contains all foods, including meat, poultry, fish and shellfish, eggs, and dairy, in addition to plant-based foods, such as fruits, vegetables, whole grains, and legumes/beans. However, red meat is limited to one time per week and poultry is limited to 5 times per week or less. We will also ask you to keep foods low in fat and low in glycemic index.
  Interventions: Behavioral: Diet
- Omnivorous (Active Comparator): An omnivorous diet contains all food groups. However, as part of this study, we will ask participants in this group to keep foods low in fat and low in glycemic index. Participants in this group will not need to attend weekly meetings but will receive information via e-mail each week.
  Interventions: Behavioral: Diet

INTERVENTIONS:
Behavioral: Diet — Change in dietary intake

SUMMARY:
Several studies have shown differences in health-related outcomes by dietary pattern. These patterns have included those participants following vegan (no meat, poultry, fish, dairy, or eggs), vegetarian (no meat, poultry, or fish), pesco- vegetarian (no meat or poultry), semi-vegetarian (red meat and poultry ≥ 1 time/month and < 1 time/week), or omnivorous diets. These studies have shown that of these dietary patterns, vegans have the lowest BMIs, lowest prevalence of Type 2 diabetes, and lowest amount of weight gain over 5 years. In addition, vegetarians have significantly better metabolic risk factors as compared to non-vegetarians. While these initial observational studies have shown benefits to consuming more plant-based diets, there have been no randomized trials examining the differences in health outcomes among these dietary patterns. To begin exploring this research area, the investigators will conduct a pilot study which will randomize participants to one of the 5 dietary approaches. Participants (n=75) in the NEW DIETs Study will be recruited to follow their randomly assigned diet for 8 weeks and attend weekly sessions to learn about nutrition and cooking.

DETAILED DESCRIPTION:
This study involves five groups. Participants will be randomly assigned to one of these groups. All groups will receive information on a dietary approach aimed at losing weight. All groups will be asked to favor foods that are low fat and have a low glycemic index, which means they will be asked to favor foods that don't cause a quick rise in blood sugar (for example, choosing oatmeal over cornflakes for breakfast). All groups will also be asked to take a vitamin B-12 supplement each day of their choosing (can be a multivitamin).

Participants who are eligible on the online screener will be contacted by phone to complete a few additional screening questions and invited to an orientation meeting.

Below are the steps in the study:

* If participants are accepted into the study, participants will come to the study site (USC Public Health Research Center) to learn more about the study, have their weight and height measured, learn how to complete questionnaires online, and complete their consent form. This meeting will last approximately 1.5 hours.
* Participants will then complete some questionnaires that measure their diet and physical activity levels on a computer at home or other location where participants have computer/internet access. We will also ask participants to keep all their grocery and restaurant receipts during this time to bring back with participants to the next meeting.
* Participants will come back for a meeting to have their weight measured again and participants will find out their diet group assignment. Participants will receive a 1.25 hour overview of the diet participants have been assigned to and be provided with materials on this diet.
* If participants are assigned to the vegan, vegetarians, pesco-, or semi-vegetarian diets, they will complete the following over the 8-week study:

  1. Participants will attend weekly meetings over 8 weeks.
  2. We will obtain their weight and collect online questionnaires at weeks 4 and 8.
  3. During the 8-week study, we will ask participants to complete an online weekly questionnaire which will assess if participants are following the diet and their weight. This will take approximately 5 minutes to complete.
* If participants are assigned to the omnivorous diet, they will only come in for meetings at baseline, 4 weeks, and 8 weeks.

  1. We will obtain their weight and collect online questionnaires at weeks 4 and 8.
  2. Participants will receive e-mailed lessons of their diet plan each week.
  3. During the 8-week study, we will ask participants to complete an online weekly questionnaire which will assess if participants are following the diet, and their weight. This will take approximately 5 minutes to complete.
  4. At week 8, participants will also be provided with information about the other 4 diets in case participants would like to try these dietary patterns after the study.
* All diet groups will be asked to collect and turn in all grocery store and restaurant receipts for 2 weeks prior to the start of the intervention and for the 8 weeks during the study.
* At study completion (8 weeks), participants will receive an incentive for participating ($20).
* Participants in all groups will be asked to take a daily multivitamin (or other reliable source of vitamin B-12) over the course of the study. You are responsible for choosing and purchasing this.
* During the study, we will ask you to keep your physical activity levels constant (keep your levels the same as what you were doing at study entry).

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 18-65
* have access to a computer with Internet capabilities
* be overweight (Body Mass Index of 25-49.9)
* be able to attend weekly evening meetings at the University of South Carolina in Columbia, SC (up to 8 total) starting late January 2013.

Exclusion Criteria: Participants will be ineligible to participate if they:

* have a Body Mass Index less than 25 or greater than 49.9 kg/m2
* are currently pregnant
* are younger than 18 or older than 65 years of age
* are unable to attend weekly meetings for 8 weeks
* don't have access to the Internet and a computer
* don't have access to a scale for self-monitoring weight
* aren't willing to be randomized to one of five dietary groups
* have a psychiatric disease, drug or alcohol dependency, or uncontrolled thyroid condition
* have a major health condition, such as heart conditions, diabetes, and past incidence of stroke
* have an eating disorder (participants will be screened using the Eating Attitudes Test screener-participants who do not pass this screener will be asked to contact their physician)
* currently participating in a weight loss program or taking weight loss medications
* currently following a vegan, vegetarian, or pesco-vegetarian diet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2012-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 8 weeks

SECONDARY OUTCOMES:
Dietary Intake | 8 weeks
  Changes in dietary intake will be measured using 2 days of 24-hour dietary recalls

CONTACTS AND LOCATIONS:
Overall Officials: Brie Turner-McGrievy, PhD, MS, RD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

REFERENCES:
- [Derived] Turner-McGrievy GM, Wirth MD, Shivappa N, Wingard EE, Fayad R, Wilcox S, Frongillo EA, Hebert JR. Randomization to plant-based dietary approaches leads to larger short-term improvements in Dietary Inflammatory Index scores and macronutrient intake compared with diets that contain meat. Nutr Res. 2015 Feb;35(2):97-106. doi: 10.1016/j.nutres.2014.11.007. Epub 2014 Dec 3. PMID 25532675